CLINICAL TRIAL: NCT07128147
Title: Detection of Helicopacter Pylori in Patients With Metabolic Associated Fatty Liver Disease
Acronym: HpyloriMAFLD
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Mohammed Abdel Mowgod, Lecturer, Tropical Medicine, Assiut University
Other Study IDs: 4-2025-300645
Record Dates: First submitted 2025-07-27; First posted 2025-08-17 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-07

CONDITIONS: Helicobacter Pylori Infection Metabolic Dysfunction-Associated Fatty Liver Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Owing to the correlation between H.pylori and MAFLD, our study aims to search for H.pylori in every patient with MAFLD to aid in the management of MAFLD and improve quality of life for these patients by decreaseing morbidity and mortality.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) has become increasingly common in recent years. NAFLD is considered the primary cause of chronic liver disorders and has emerged as a significant global public health concern.

The prevalence of NAFLD has been steadily rising due to changes in lifestyle and dietary habits, making it the most common chronic liver disease worldwide. The global prevalence of NAFLD is estimated at 30.1%.

Recently, researchers published an international expert consensus statement introducing a new definition: metabolic dysfunction-associated fatty liver disease (MAFLD), intended to replace the term non-alcoholic fatty liver disease (NAFLD).

The new nomenclature, MAFLD, is based on the presence of steatosis in more than 5% of hepatocytes, along with the absence of excessive alcohol consumption or other causes of chronic liver disease. A diagnosis of MAFLD can be established by the presence of hepatic steatosis in combination with one of the following three criteria: overweight/obesity, type 2 diabetes mellitus, or evidence of metabolic dysregulation.

Metabolic dysregulation is defined as having at least two of the following metabolic risk abnormalities: increased waist circumference, elevated blood pressure, dyslipidemia, prediabetes, insulin resistance, or elevated plasma C-reactive protein levels.

One potential hidden cause of cryptogenic cirrhosis is "burned-out" NAFLD. Therefore, early treatment of NAFLD and its underlying risk factors is crucial to prevent liver damage and potential liver failure.

Research has shown that abnormal lipid metabolism in the liver can lead to dysbiosis of the intestinal flora. This imbalance can further promote lipid accumulation in the liver. Additionally, NAFLD has been associated with gut microbiota alterations, particularly involving Helicobacter pylori (H. pylori).

Globally, infection with H. pylori affects approximately 50% or more of the population. H. pylori is a gram-negative bacterium that colonizes the human stomach and is known for its role in various gastrointestinal diseases. It is a major etiological factor in chronic peptic ulcer disease, which includes both gastric and duodenal ulcers.

The bacterium's ability to survive in the stomach's acidic environment is facilitated by its production of urease, an enzyme that neutralizes stomach acid. Chronic H. pylori infection can result in complications such as peptic ulcers, gastritis, and chronic indigestion (dyspepsia), making it a significant global public health issue. It may also lead to serious conditions like gastric adenocarcinoma and mucosa-associated lymphoid tissue (MALT) lymphoma.

Furthermore, some researchers have found a connection between H. pylori and liver cancer, diabetes, and disrupted lipid metabolism.

Several studies have indicated that H. pylori infection is one of the contributing factors in the progression of NAFLD and that eradication of H. pylori may partially halt the development of the disease.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged >18 years old.
* Was diagnosed as MAFLD based on abdominal ultrasonography (US) or other imaging techniques.

Exclusion Criteria:

* Patients aged ≤18 years old.
* Pregnancy.
* Presence of malignancy.
* Type I DM.
* Patients with fatty liver who undergone bariatric surgeries.
* Previous history of alcohol consumption, steroids, proton pump inhibitors, antibiotics, and contraceptive pills.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients, and their relatives, were invited to do screening for fatty liver by doing conventional abdominal ultrasound (US) by any member of the nutrition clinic team for assessment of liver echopattern.Patients with detected bright liver by US suggestive of fatty liver have undergone an evaluation for the BMI and tests to detect metabolic risk abnormalities.Diagnosis of MAFLD was made when a patient has BMI >25 kg/m2, T2DM or at least two metabolic risk abnormalities.Our study will use either H.pylori stool antigen test (SAT), after stoppage of PPI and antibiotics two weeks before the test, as it cheap and easy, or diagnostic upper endoscopy with biopsy.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Helicobacter pylori infection in patients with Metabolic Associated Fatty Liver Disease as determined by Urea Breath Test | Baseline (Day 1 of hospital admission)
  H. pylori infection will be assessed at baseline using a standardized H.pylori antigen in stool. Results will be reported as the proportion (%) of patients with a positive test among all enrolled participants
Prevalence of Helicobacter pylori Infection in Patients with MAFLD | At baseline (hospital admission)
  Detection of H. pylori infection using [stool antigen test /endoscopic biopsy] in patients diagnosed with MAFLD

CONTACTS AND LOCATIONS:
Overall Officials: Amira M Assiut University, Lecturer, MD, Trop Med, Principal Investigator — Assiut University